CLINICAL TRIAL: NCT01864447
Title: An Exercise Training and Behavioral Weight Loss Program After an Acute Blood Clot: TRAIN ABC
Brief Title: Exercise Training After an Acute Blood Clot
Acronym: TRAIN ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Susan Lakoski, Assistant Professor, University of Vermont College of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS M13-219
Record Dates: First submitted 2013-05-17; First posted 2013-05-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: VTE
Keywords: VTE; Exercise; Diet; Weight loss; DVT; PE
MeSH Terms: conditions — Motor Activity; Weight Loss | interventions — HCE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VTE REHABILITATION (Experimental): The exercise prescription emphasizes gradual progression to longer duration (45-60 minutes per session), lower intensity (60-70% peak heart rate (PHR) exercise. Subjects have an exercise expenditure goal of >3000 kcal/wk, attained after 2 to 4 weeks of gradually lengthening exercise bouts. All exercise sessions will be performed onsite for the first two weeks, after which subjects will perform 2 additional sessions a week in the home environment. Exercise logs will be reviewed weekly.
  The Dietary Behavioral Weight Loss Intervention(BWL) intervention consists primarily of 12 small group sessions led by a dietician emphasizing dietary records, itemization of food, and caloric content. Subjects will be given individualized daily caloric goals 500 kcal less than predicted maintenance calories based on their baseline body weight.
  Interventions: Behavioral: VTE REHABILITATION: High-Caloric Expenditure Exercise Training (HCE) and The Dietary Behavioral Weight Loss Intervention (BWL)
- CONTROL (No Intervention): The 12-week program will consist of monthly phone contacts to check-in to capture physical activity done outside of the intervention setting.

INTERVENTIONS:
Behavioral: VTE REHABILITATION: High-Caloric Expenditure Exercise Training (HCE) and The Dietary Behavioral Weight Loss Intervention (BWL)
  Arms: VTE REHABILITATION

SUMMARY:
Patients after an acute blood clot in the veins are at risk for leg-related complications such as pain, swelling, and immobility. In addition, the occurrence of blood clots can have major implications for personal health including weight gain, blood clot recurrence and impairment in cardiovascular functioning. The goal of this study is to determine whether aerobic exercise training is a therapeutic strategy to offset risk factors for recurrent blood clots or leg complications.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR), a formalized exercise and behavioral modification program, is the cornerstone of secondary prevention for heart disease. Implementation of CR early after an acute myocardial infarction (MI) is associated with improved cardiac function and survival. As such, CR is now standard of care for a majority of hospital-based discharge programs following coronary events. In stark contrast, no similar program exists following an acute venous thromboembolism (VTE or blood clot), despite a high rate of limb and respiratory disability after VTE, shared risk factors with heart disease, and known beneficial impact of exercise training on VTE complications (e.g. post-thrombotic syndrome, PTS).

Body weight is a key modifiable risk factor driving risk of incident and recurrent VTE. Obese patients with prior VTE have a 2-fold higher risk of a second VTE compared to normal weight patients.(1) Importantly, VTE recurrence risk escalates if weight control is not established. Weight gain after acute DVT is common, with a mean 7% increase over 6 months.(2) To date, however, there is limited evidence regarding whether early initiation of exercise training following acute DVT is safe and feasible and mitigates weight gain associated with a VTE diagnosis. Previously, a significant decrease in body weight and fat mass loss was demonstrated utilizing high-caloric expenditure exercise in the CR setting.(3) Delineating the impact of high-caloric expenditure exercise to induce weight loss and reduce VTE complications and recurrence is a critical first step toward evaluating the role of early post-VTE rehabilitation in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute unprovoked proximal or distal DVT >= 6 weeks
* On anticoagulation therapy
* Patient self-report of ability to walk 10 minutes without interruption or pain
* Age >=16 and <80
* Willingness to participate in exercise rehabilitation program at Tilley Drive South Burlington

Exclusion Criteria:

* Symptomatic PE, defined as 1) right heart strain as assessed by computed tomography or echocardiogram, 2) resting hypoxia - resting oxygen saturation <92%
* Provoked VTE: major surgery, trauma, or pregnancy
* Medical condition that alters ability to walk for exercise

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Obesity and VTE Recurrence | 3 months
  Blood work will be taken at baseline and 3 months. Measures will include adiponectin, leptin, resistin, visfatin, CRP, IL-6, PAI-1, endogenous thrombin potential, and D-dimer.Samples will be processed in the clinic with attention to issues related to coagulation activation, and plasma and serum will be stored at -80 degrees C in our laboratory.

SECONDARY OUTCOMES:
Maximal Exercise Capacity | 3 months
  Maximal exercise capacity will be assessed on the treadmill with measurement of peak oxygen uptake, duration of treadmill exercise and maximal exercise intensity in METS. A continuous modified-Balke protocol will be used, with exercise increasing gradually at 1 MET increments at 2 minute intervals.

OTHER OUTCOMES:
Feasibility | 3 months
  Feasibility will be evaluated by assessing the rates of study eligibility, acceptance, and overall accrual.
Safety | every 4 weeks, for up to 12 weeks
  Safety will be evaluated by the type and prevalence of adverse events during exercise-related assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Susan G Lakoski, MD, Principal Investigator — University of Vermont
Locations (1):
- Flether Allen Healthcare, Burlington, Vermont, United States

REFERENCES:
- [Background] Eichinger S, Hron G, Bialonczyk C, Hirschl M, Minar E, Wagner O, Heinze G, Kyrle PA. Overweight, obesity, and the risk of recurrent venous thromboembolism. Arch Intern Med. 2008 Aug 11;168(15):1678-83. doi: 10.1001/archinte.168.15.1678. PMID 18695082
- [Background] Ageno W, Piantanida E, Dentali F, Mera V, Squizzato A, Marchesi C, Steidl L, Venco A. Weight gain after acute deep venous thrombosis: a prospective observational study. Thromb Res. 2003 Jan 1;109(1):31-5. doi: 10.1016/s0049-3848(03)00145-2. PMID 12679129
- [Background] Ades PA, Savage PD, Toth MJ, Harvey-Berino J, Schneider DJ, Bunn JY, Audelin MC, Ludlow M. High-calorie-expenditure exercise: a new approach to cardiac rehabilitation for overweight coronary patients. Circulation. 2009 May 26;119(20):2671-8. doi: 10.1161/CIRCULATIONAHA.108.834184. Epub 2009 May 11. PMID 19433757
- [Background] Hirsh J, Hoak J. Management of deep vein thrombosis and pulmonary embolism. A statement for healthcare professionals. Council on Thrombosis (in consultation with the Council on Cardiovascular Radiology), American Heart Association. Circulation. 1996 Jun 15;93(12):2212-45. doi: 10.1161/01.cir.93.12.2212. No abstract available. PMID 8925592
- [Background] Heit JA, Mohr DN, Silverstein MD, Petterson TM, O'Fallon WM, Melton LJ 3rd. Predictors of recurrence after deep vein thrombosis and pulmonary embolism: a population-based cohort study. Arch Intern Med. 2000 Mar 27;160(6):761-8. doi: 10.1001/archinte.160.6.761. PMID 10737275
- [Background] Prandoni P, Lensing AW, Cogo A, Cuppini S, Villalta S, Carta M, Cattelan AM, Polistena P, Bernardi E, Prins MH. The long-term clinical course of acute deep venous thrombosis. Ann Intern Med. 1996 Jul 1;125(1):1-7. doi: 10.7326/0003-4819-125-1-199607010-00001. PMID 8644983
- [Background] Carrier M, Le Gal G, Wells PS, Rodger MA. Systematic review: case-fatality rates of recurrent venous thromboembolism and major bleeding events among patients treated for venous thromboembolism. Ann Intern Med. 2010 May 4;152(9):578-89. doi: 10.7326/0003-4819-152-9-201005040-00008. PMID 20439576
- [Background] Douketis JD, Gu CS, Schulman S, Ghirarduzzi A, Pengo V, Prandoni P. The risk for fatal pulmonary embolism after discontinuing anticoagulant therapy for venous thromboembolism. Ann Intern Med. 2007 Dec 4;147(11):766-74. doi: 10.7326/0003-4819-147-11-200712040-00007. PMID 18056660
- [Background] Ageno W, Becattini C, Brighton T, Selby R, Kamphuisen PW. Cardiovascular risk factors and venous thromboembolism: a meta-analysis. Circulation. 2008 Jan 1;117(1):93-102. doi: 10.1161/CIRCULATIONAHA.107.709204. Epub 2007 Dec 17. PMID 18086925
- [Background] Kahn SR, Shrier I, Julian JA, Ducruet T, Arsenault L, Miron MJ, Roussin A, Desmarais S, Joyal F, Kassis J, Solymoss S, Desjardins L, Lamping DL, Johri M, Ginsberg JS. Determinants and time course of the postthrombotic syndrome after acute deep venous thrombosis. Ann Intern Med. 2008 Nov 18;149(10):698-707. doi: 10.7326/0003-4819-149-10-200811180-00004. PMID 19017588
- [Background] Barlow CE, Defina LF, Radford NB, Berry JD, Cooper KH, Haskell WL, Jones LW, Lakoski SG. Cardiorespiratory fitness and long-term survival in "low-risk" adults. J Am Heart Assoc. 2012 Aug;1(4):e001354. doi: 10.1161/JAHA.112.001354. Epub 2012 Aug 24. PMID 23130161
- [Background] Berry JD, Willis B, Gupta S, Barlow CE, Lakoski SG, Khera A, Rohatgi A, de Lemos JA, Haskell W, Lloyd-Jones DM. Lifetime risks for cardiovascular disease mortality by cardiorespiratory fitness levels measured at ages 45, 55, and 65 years in men. The Cooper Center Longitudinal Study. J Am Coll Cardiol. 2011 Apr 12;57(15):1604-10. doi: 10.1016/j.jacc.2010.10.056. PMID 21474041
- [Background] Gupta S, Rohatgi A, Ayers CR, Willis BL, Haskell WL, Khera A, Drazner MH, de Lemos JA, Berry JD. Cardiorespiratory fitness and classification of risk of cardiovascular disease mortality. Circulation. 2011 Apr 5;123(13):1377-83. doi: 10.1161/CIRCULATIONAHA.110.003236. Epub 2011 Mar 21. PMID 21422392
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Belardinelli R, Georgiou D, Cianci G, Purcaro A. 10-year exercise training in chronic heart failure: a randomized controlled trial. J Am Coll Cardiol. 2012 Oct 16;60(16):1521-8. doi: 10.1016/j.jacc.2012.06.036. Epub 2012 Sep 19. PMID 22999730
- [Background] Sierra-Johnson J, Romero-Corral A, Somers VK, Lopez-Jimenez F, Thomas RJ, Squires RW, Allison TG. Prognostic importance of weight loss in patients with coronary heart disease regardless of initial body mass index. Eur J Cardiovasc Prev Rehabil. 2008 Jun;15(3):336-40. doi: 10.1097/HJR.0b013e3282f48348. PMID 18525390
- [Background] Blattler W, Partsch H. Leg compression and ambulation is better than bed rest for the treatment of acute deep venous thrombosis. Int Angiol. 2003 Dec;22(4):393-400. PMID 15153824
- [Background] Junger M, Diehm C, Storiko H, Hach-Wunderle V, Heidrich H, Karasch T, Ochs HR, Ranft J, Sannwald GA, Strolin A, Janssen D. Mobilization versus immobilization in the treatment of acute proximal deep venous thrombosis: a prospective, randomized, open, multicentre trial. Curr Med Res Opin. 2006 Mar;22(3):593-602. doi: 10.1185/030079906X89838. PMID 16574042
- [Background] Partsch H, Kaulich M, Mayer W. Immediate mobilisation in acute vein thrombosis reduces post-thrombotic syndrome. Int Angiol. 2004 Sep;23(3):206-12. PMID 15765034
- [Background] Kahn SR, Azoulay L, Hirsch A, Haber M, Strulovitch C, Shrier I. Acute effects of exercise in patients with previous deep venous thrombosis: impact of the postthrombotic syndrome. Chest. 2003 Feb;123(2):399-405. doi: 10.1378/chest.123.2.399. PMID 12576357
- [Background] Kahn SR, Shrier I, Shapiro S, Houweling AH, Hirsch AM, Reid RD, Kearon C, Rabhi K, Rodger MA, Kovacs MJ, Anderson DR, Wells PS. Six-month exercise training program to treat post-thrombotic syndrome: a randomized controlled two-centre trial. CMAJ. 2011 Jan 11;183(1):37-44. doi: 10.1503/cmaj.100248. Epub 2010 Nov 22. PMID 21098066
- [Background] Isma N, Johanssson E, Bjork A, Bjorgell O, Robertson F, Mattiasson I, Gottsater A, Lindblad B. Does supervised exercise after deep venous thrombosis improve recanalization of occluded vein segments? A randomized study. J Thromb Thrombolysis. 2007 Feb;23(1):25-30. doi: 10.1007/s11239-006-9010-y. PMID 17186396
- [Background] Murdolo G, Smith U. The dysregulated adipose tissue: a connecting link between insulin resistance, type 2 diabetes mellitus and atherosclerosis. Nutr Metab Cardiovasc Dis. 2006 Mar;16 Suppl 1:S35-8. doi: 10.1016/j.numecd.2005.10.016. Epub 2006 Feb 9. PMID 16530128
- [Background] Rosito GA, D'Agostino RB, Massaro J, Lipinska I, Mittleman MA, Sutherland P, Wilson PW, Levy D, Muller JE, Tofler GH. Association between obesity and a prothrombotic state: the Framingham Offspring Study. Thromb Haemost. 2004 Apr;91(4):683-9. doi: 10.1160/th03-01-0014. PMID 15045128
- [Background] Folsom AR, Qamhieh HT, Wing RR, Jeffery RW, Stinson VL, Kuller LH, Wu KK. Impact of weight loss on plasminogen activator inhibitor (PAI-1), factor VII, and other hemostatic factors in moderately overweight adults. Arterioscler Thromb. 1993 Feb;13(2):162-9. doi: 10.1161/01.atv.13.2.162. PMID 8427853
- [Background] Loskutoff DJ, Samad F. The adipocyte and hemostatic balance in obesity: studies of PAI-1. Arterioscler Thromb Vasc Biol. 1998 Jan;18(1):1-6. doi: 10.1161/01.atv.18.1.1. No abstract available. PMID 9445248
- [Background] Marckmann P, Toubro S, Astrup A. Sustained improvement in blood lipids, coagulation, and fibrinolysis after major weight loss in obese subjects. Eur J Clin Nutr. 1998 May;52(5):329-33. doi: 10.1038/sj.ejcn.1600558. PMID 9630382
- [Background] Alessi MC, Morange P, Juhan-Vague I. Fat cell function and fibrinolysis. Horm Metab Res. 2000 Nov-Dec;32(11-12):504-8. doi: 10.1055/s-2007-978677. PMID 11246816
- [Background] Shi Y, Tokunaga O. Chlamydia pneumoniae (C. pneumoniae) infection upregulates atherosclerosis-related gene expression in human umbilical vein endothelial cells (HUVECs). Atherosclerosis. 2004 Dec;177(2):245-53. doi: 10.1016/j.atherosclerosis.2004.07.014. PMID 15530896
- [Background] Soderberg S, Olsson T, Eliasson M, Johnson O, Ahren B. Plasma leptin levels are associated with abnormal fibrinolysis in men and postmenopausal women. J Intern Med. 1999 May;245(5):533-43. doi: 10.1046/j.1365-2796.1999.00472.x. PMID 10363755
- [Background] Skurk T, van Harmelen V, Lee YM, Wirth A, Hauner H. Relationship between IL-6, leptin and adiponectin and variables of fibrinolysis in overweight and obese hypertensive patients. Horm Metab Res. 2002 Nov-Dec;34(11-12):659-63. doi: 10.1055/s-2002-38253. PMID 12660878
- [Background] Beltowski J. Leptin and atherosclerosis. Atherosclerosis. 2006 Nov;189(1):47-60. doi: 10.1016/j.atherosclerosis.2006.03.003. Epub 2006 Apr 3. PMID 16580676
- [Background] Allison MA, Cushman M, Callas PW, Denenberg JO, Jensky NE, Criqui MH. Adipokines are associated with lower extremity venous disease: the San Diego population study. J Thromb Haemost. 2010 Sep;8(9):1912-8. doi: 10.1111/j.1538-7836.2010.03941.x. PMID 20546124
- [Background] D'Zurilla TJ, Goldfried MR. Problem solving and behavior modification. J Abnorm Psychol. 1971 Aug;78(1):107-26. doi: 10.1037/h0031360. No abstract available. PMID 4938262
- [Background] Green D. Risk of future arterial cardiovascular events in patients with idiopathic venous thromboembolism. Hematology Am Soc Hematol Educ Program. 2009:259-66. doi: 10.1182/asheducation-2009.1.259. PMID 20008208
- [Background] Kahn SR. Measurement properties of the Villalta scale to define and classify the severity of the post-thrombotic syndrome. J Thromb Haemost. 2009 May;7(5):884-8. doi: 10.1111/j.1538-7836.2009.03339.x. Epub 2009 Mar 6. PMID 19320818
- [Background] Kahn SR, Desmarais S, Ducruet T, Arsenault L, Ginsberg JS. Comparison of the Villalta and Ginsberg clinical scales to diagnose the post-thrombotic syndrome: correlation with patient-reported disease burden and venous valvular reflux. J Thromb Haemost. 2006 Apr;4(4):907-8. doi: 10.1111/j.1538-7836.2006.01824.x. No abstract available. PMID 16634767
- [Background] Kahn SR, Lamping DL, Ducruet T, Arsenault L, Miron MJ, Roussin A, Desmarais S, Joyal F, Kassis J, Solymoss S, Desjardins L, Johri M, Shrier I; VETO Study investigators. VEINES-QOL/Sym questionnaire was a reliable and valid disease-specific quality of life measure for deep venous thrombosis. J Clin Epidemiol. 2006 Oct;59(10):1049-56. doi: 10.1016/j.jclinepi.2005.10.016. Epub 2006 Jun 23. PMID 16980144